CLINICAL TRIAL: NCT04332380
Title: Convalescent Plasma for Patients With COVID-19: A Pilot Study
Acronym: CP-COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universidad del Rosario (Other)
Collaborators: CES University (Other); Instituto Distrital de Ciencia Biotecnologia e Innovacion en salud (Unknown); Fundación Universitaria de Ciencias de la Salud (Other)
Responsible Party: Principal Investigator, Juan Manuel Anaya Cabrera, MD, PhD, Principal Investigator, Universidad del Rosario
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABN011-1
Record Dates: First submitted 2020-03-30; First posted 2020-04-02 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Coronavirus; Coronavirus Infection
Keywords: COVID-19; Coronavirus Disease 2019
MeSH Terms: conditions — Coronavirus Infections; COVID-19 | interventions — COVID-19 Serotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): Participants included in the experimental group will receive 500 milliliters of convalescent plasma, distributed in two 250 milliliters transfusions on the first and second day after starting the protocol.
  Interventions: Drug: Plasma

INTERVENTIONS:
Drug: Plasma — Day 1: CP-COVID19, 250 milliliters. Day 2: CP-COVID19, 250 milliliters.
  Other Names: Convalescent Plasma COVID-19

SUMMARY:
Convalescent plasma (CP) has been used in recent years as an empirical treatment strategy when there is no vaccine or treatment available for infectious diseases. In the latest viral epidemics, such as the Ebola outbreak in West Africa in 2014, the World Health Organization issued a document outlining a protocol for the use of whole blood or plasma collected from patients who have recovered from the Ebola virus disease by transfusion to empirically treat local infectious outbreaks.

DETAILED DESCRIPTION:
The process is based on obtaining plasma from patients recovered from COVID-19 in Colombia, and through a donation of plasma from the recovered, the subsequent transfusion of this to patients infected with coronavirus disease (COVID-19). Our group has reviewed the scientific evidence regarding the application of convalescent plasma for emergency viral outbreaks and has recommended the following protocol

ELIGIBILITY:
Inclusion Criteria:Fulfilling all the following criteria

1. Aged between 18 and 60 years, male or female.
2. Hospitalized participants with diagnosis for COVID 19 by Real Time - Polymerase Chain Reaction.
3. Without treatment.
4. Moderate cases according to the official guideline "Pneumonia Diagnosis and Treatment Scheme for Novel Coronavirus Infection (Trial Version 6)".
5. Confusion, Urea, Respiratory rate, Blood pressure-65 (CURB-65) >= 2.
6. Sequential Organ Failure Assessment score (SOFA) < 6.
7. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Female subjects who are pregnant or breastfeeding.
2. Patients with prior allergic reactions to transfusions.
3. Critical ill patients in intensive care units.
4. Patients with surgical procedures in the last 30 days.
5. Patients with active treatment for cancer (Radiotherapy or Chemotherapy).
6. HIV diagnosed patients with viral failure (detectable viral load> 1000 copies / ml persistent, two consecutive viral load measurements within a 3 month interval, with medication adherence between measurements after at least 6 months of starting a new regimen antiretrovirals).
7. Patients who have suspicion or evidence of coinfections.
8. End-stage chronic kidney disease (Glomerular Filtration Rate <15 ml / min / 1.73 m2).
9. Child Pugh C stage liver cirrhosis.
10. High cardiac output diseases.
11. Autoimmune diseases or Immunoglobulin A nephropathy.
12. Patients have any condition that in the judgement of the Investigators would make the subject inappropriate for entry into this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-07-28 (Actual); Study Completion 2020-07-28 (Actual)

PRIMARY OUTCOMES:
Change in Viral Load | Days 0, 4, 7, 14 and 28
  Copies of COVID-19 per ml
Change in Immunoglobulin M COVID-19 antibodies Titers | Days 0, 4, 7, 14 and 28
  Immunoglobulin M COVID-19 antibodies
Change in Immunoglobulin G COVID-19 antibodies Titers | Days 0, 4, 7, 14 and 28
  Immunoglobulin G COVID-19 antibodies

SECONDARY OUTCOMES:
Intensive Care Unit Admission | Days 7, 14 and 28
  Proportion of patients with Intensive Care Unit Admission requirement (days 7, 14 and 28)
Length of Intensive Care Unit stay | Days 7, 14 and 28
  Days of Intensive Care Unit management (days 7, 14 and 28)
Length of hospital stay (days) | Days 7, 14 and 28
  Days of Hospitalization (days 7, 14 and 28)
Requirement of mechanical ventilation | Days 7, 14 and 28
  Proportion of patients with mechanical ventilation (days 7, 14 and 28)
Duration (days) of mechanical ventilation | Days 7, 14 and 28
  Days with mechanical ventilation (days 7, 14 and 28)
Clinical status assessed according to the World Health Organization guideline | Days 7, 14 and 28
  1. Hospital discharge; 2. Hospitalization, not requiring supplemental oxygen; 3. Hospitalization, requiring supplemental oxygen (but not Noninvasive Ventilation/ HFNC); 4. Intensive care unit/hospitalization, requiring Noninvasive Ventilation/ HFNC therapy; 5. Intensive care unit, requiring extracorporeal membrane oxygenation and/or invasive mechanical ventilation; 6. Death. (days 7, 14 and 28)
Mortality | Days 7, 14 and 28
  Proportión of death patients at days 7, 14 and 28

CONTACTS AND LOCATIONS:
Overall Officials: Juan M Anaya Cabrera, MD, PhD, Principal Investigator — Universidad del Rosario
Locations (1):
- Universidad del Rosario, Bogota, Cundinamarca, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Wang Y, Wang Y, Chen Y, Qin Q. Unique epidemiological and clinical features of the emerging 2019 novel coronavirus pneumonia (COVID-19) implicate special control measures. J Med Virol. 2020 Jun;92(6):568-576. doi: 10.1002/jmv.25748. Epub 2020 Mar 29. PMID 32134116
- [Background] Young BE, Ong SWX, Kalimuddin S, Low JG, Tan SY, Loh J, Ng OT, Marimuthu K, Ang LW, Mak TM, Lau SK, Anderson DE, Chan KS, Tan TY, Ng TY, Cui L, Said Z, Kurupatham L, Chen MI, Chan M, Vasoo S, Wang LF, Tan BH, Lin RTP, Lee VJM, Leo YS, Lye DC; Singapore 2019 Novel Coronavirus Outbreak Research Team. Epidemiologic Features and Clinical Course of Patients Infected With SARS-CoV-2 in Singapore. JAMA. 2020 Apr 21;323(15):1488-1494. doi: 10.1001/jama.2020.3204. PMID 32125362
- [Background] Infectious, D. & Outbreaks, D. Maintaining a safe and adequate blood supply during the pandemic outbreak of coronavirus disease ( COVID-19 ). OMS 1-5 (2020).